# A Randomized Trial of Social and Financial Incentives to Increase Physical Activity Among Overweight and Obese Veterans

NCT# 03563027

April 17, 2020

## Analysis Implementation Plan - VA Study Trial

#### 1. Data Checks

a. For each variable (outcome and characteristics/predictor) calculate the following percentiles: 1, 5, 10, 25, 50, 75, 90, 95, 99

#### 2. Missing Data

- a. For outcome variables (Daily Steps) identify missing values at weeks 1-12, 1-4, 5-12, and 13-20
- b. For Steps separately list values that are missing from values that are <1000

## 3. Participant characteristics

- a. Create Table 1
- b. Estimate baseline measures

### 4. Imputation plan

- a. Change in mean daily steps
  - Model driven approach to run 5 imputations for any missing values or values < 1000 steps</li>
  - ii. Covariates include: study arm, week of study, calendar month, baseline step count, age, gender, race/ethnicity, education, marital status, annual household income, military service period, and BMI

#### 5. Unadjusted: Estimate Mean and SD for outcome measures (using imputed data)

- a. Daily steps during baseline, weeks 5-12, weeks 13-20 and weeks 1-20
  - i. Graph monthly trends
- b. Proportion of days achieving step goal during 5-12 weeks and weeks 13-20

## 6. Adjusted changes in outcome measures (imputed model is primary; non-imputed is secondary)

- a. Use generalized linear mixed models (GLIMMIX) with identity link for mean change in daily steps during weeks 5-12 and weeks 13-20.
  - i. Adjusted for baseline steps, calendar month, study arm, participant random effect
- b. Use generalized linear mixed models (GLIMMIX) with logit link (logistic model) for proportion of days achieving step goal during weeks 5-12 and weeks 13-20
  - i. Adjusted for baseline steps, calendar month, study arm, participant random effect
  - ii. Use 1000 bootstrapped samples to find adjusted changes in percentage points with 95% confidence intervals for proportion of days achieving step goals

#### 7. Survey Measures

a. Tech access and use, IPAQ, follow-up survey